CLINICAL TRIAL: NCT07017166
Title: Development of a Clinical Screening, Diagnostic and Evaluation Tool for Patients With Lower Limb Lymphedema (LLL): To Develop an Evaluation Set for Patients With LLL (AIM 5)
Brief Title: Development of a Clinical Screening, Diagnostic and Evaluation Tool for Patients With Lower Limb Lymphedema: Aim 5
Acronym: EvaLymph-Leg5
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S66033-aim5
Record Dates: First submitted 2025-06-02; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-05

CONDITIONS: Lower Limb Lymphedema
Keywords: Lymphedema; Measurement; Clinical evaluation; Reliability; Validity; Lower limb; Structure sensor scanner
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 33 patients with LLL: patients with unilateral or bilateral, primary or secundary LLL who visit the center for lymphedema at UZ Leuven

SUMMARY:
This clinical study evaluates the reliability, concurrent validity, and clinical feasibility of a new method to determine leg volume, namely the Structure Sensor Scanner.

The volume of both legs will be determined using three different measurement methods:

1. A scanning method using a Structure Sensor Scanner: for this, both legs are scanned all around with an iPad with the Structure Sensor attached to the tablet. This is performed while standing. The sensor captures depth images, which are then converted into a three-dimensional image of both legs. A computer program is then used to determine the volume of both legs and specific segments of the legs.
2. The circumference measurement using a perimeter: the perimeter consists of a flexible metal strip with a tape measure attached every 4 cm, each ending in a small weight. The person must sit and place only the foot on a small bench so that the entire leg is free. The perimeter is then placed on the leg. Finally, the tape measures are wrapped around the leg, and the circumferences are read. The leg volume is then calculated using the formula of the truncated cone.
3. The optoelectronic volumetry using the Perometer®: for this, the person must stand in shoulder-width stance on the Perometer platform, with one leg inside the frame. The frame is then moved upward. The frame captures silhouettes from which circumference and volumes are calculated through elliptical approximation.

To investigate the reliability, the intra-class correlation coefficient (ICC) is calculated as well as the SEM, SRD and a two-tailed paired samples t-test or a wilcoxon signed rank test (in case of not-normally distributed data). To investigate the concurrent validity of the Structure Sensor Scanner, the results from the scanner method will be compared with those of the two other methods. Regarding the clinical feasibility the duration of each measurement is recorded and a purpose-designed feasibility questionnaire which is completed by the assessors is used.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral or bilateral, primary or secondary LLL
* Objective diagnosis of lymphedema: ≥ 5% volume difference OR ≥ 2 minor/ 1 major criteria on lymphoscintigraphy OR presence of ICG dermal backflow
* Age ≥ 18 years
* Able to read, understand and speak Dutch

Exclusion Criteria:

* Pregnant participants
* Presence of chronic venous insufficiency C4, C5, C6; deep venous thrombosis; post-thrombotic syndrome
* Presence of skin infections of wounds at the level of the lower limbs at the moment of inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with unilateral or bilateral, primary or secondary LLL will be recruited at the center for lymphedema in UZ Leuven.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2024-02-20 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-03-28 (Actual)

PRIMARY OUTCOMES:
Within-session reliability of leg volume measurements using the Structure Sensor Scanner, circumference measurements, and optoelectronic volumetry. | One visit linked to a routine follow-up appointment at the hospital (within-session)
  Leg volumes were measured using three methods: the Structure Sensor Scanner device, manual circumference measurements, and optoelectronic volumetry. Intra-rater and inter-rater reliability were assessed through two measurements conducted by assessor A and one by assessor B. Reliability was evaluated using Intraclass Correlation Coefficients (ICC), Standard Error of Measurement (SEM), paired samples t-tests, and Smallest Real Difference (SRD).
Within-session concurrent validity of leg volume measurements using the Structure Sensor Scanner, circumference measurements, and optoelectronic volumetry. | One visit linked to a routine follow-up appointment at the hospital (within-session)
  Leg volumes were measured using three methods: the Structure Sensor Scanner device, manual circumference measurements, and optoelectronic volumetry. Concurrent validity was assessed through Pearson correlation coefficients between the measurement methods.
Clinical feasibility of leg volume measurements using the Structure Sensor Scanner, circumference measurements, and optoelectronic volumetry. | One visit linked to a routine follow-up appointment at the hospital
  Leg volumes were measured using three methods: the Structure Sensor Scanner device, manual circumference measurements, and optoelectronic volumetry. Clinical feasibility was determined by recording the duration of each measurement and using a purpose-designed feasibility questionnaire completed by the assessors.

CONTACTS AND LOCATIONS:
Overall Officials: Nele Devoogdt, PhD, Principal Investigator — KU Leuven
Locations (1):
- University Hospitals of Leuven, center for lymphedema, Leuven, Belgium